CLINICAL TRIAL: NCT06596200
Title: Pilot Study for the Use of Spinal Cord Stimulation to Alleviate Pain from Chemotherapy Induced Peripheral Neuropathy Due to Taxane or Platinum Based Agents
Brief Title: Spinal Cord Stimulation for Chemotherapy Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland St. Joseph Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00110894
Record Dates: First submitted 2024-07-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Group - SCS (Experimental): Patients who are eligible will receive a trial implant for a 3-7 day trial period. If there is at least 50% pain relief in the trial period, the patients will receive the permanent SCS implant and will be followed for 1 year post permanent implant.
  Interventions: Device: Spinal Cord Stimulation Implant

INTERVENTIONS:
Device: Spinal Cord Stimulation Implant — Spinal Cord Stimulation using 10 kHz stimulation to the thoracic spinal cord

SUMMARY:
Spinal Cord Stimulation using 10 kHz stimulation to the thoracic spinal cord will be a safe and effective treatment for CIPN, reducing pain in the lower extremities by at least 50%.

ELIGIBILITY:
Inclusion Criteria:

* CIPN as diagnosed by Oncology and/or neurology
* Receipt of a platinum-based or taxane chemotherapy prior to development of CIPN
* Pain severity greater than 4 out of 10 on a numeric rating scale of pain
* Pain chronicity greater than 6 months after the cessation of chemotherapy
* Failure of medical therapy, which must have included duloxetine
* Age 18 or greater

Exclusion Criteria:

* Platelet count less than 100k/mm3
* Spinal anatomy precluding placement of the SCS leads between T6 and T11
* Active infection
* Estimated Lifespan less than 1 year
* Receipt of vincristine, thalidomide, bortezomib, or eribulin within the prior 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
-- Measure response of CIPN pain to HF10 treatment using the numeric scale of pain (NRS) at SCS trial for all subjects and at 3, 6 and 12 months after implant for subjects who qualify for permanent implant. | 1 year

SECONDARY OUTCOMES:
- - Neuropathy symptoms will be quantified using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale (CIPN20). CIPN20 is a 20-item patient questionnaire with items scored 1 to 4. | 1 year
  CIPN20 is a 20-item patient questionnaire with items scored 1 to 4. Scores vary from 20 to 80, with higher scores indicating more prevalent neuropathy symptoms.
- Pain interference in daily life will be quantified via the brief pain inventory (BPI). | 1 year
  BPI includes reported pain severity (NRS) and a 7-item questionnaire assessing pain interference with each item scored 0-10 with higher scores indicating worsened pain interference.
- Neuropathy findings will be quantified with the modified Toronto clinical neuropathy score (mTCNS). | 1 year
  The mTCNS is a clinician administered exam with 11 items scored 0-3. A normal score is 0 with higher scores indicating worsened neuropathy on physical exam, up to a maximum of 33.
- The subject's impression of SCS efficacy will be measured using the patient global impression of change (PGIC). | 1 year
  PGIC is a 7 point scale rating their impression (1-"very much improved", 2-"much improved", 3-"minimally improved", 4-"no change", 5-"minimally worse", 6-"much worse", 7-"very much worse").
- Health related quality of life will be assessed using the EuroQOL5D-5L questionnaire. | 1 year
- Any treatment related adverse events observed during the trial will be documented using the Common Terminology Criteria for Adverse Events (CTCAE) ver 5.0. | 1 year

IPD SHARING:
Plan to Share IPD: No